CLINICAL TRIAL: NCT02834117
Title: Comparison of the Number of Visits and the Quality of Life Versus Natural Cycle in Stimulated Cycle Before Frozen Embryo Transfer
Brief Title: Natural Cycle Versus Stimulated Cycle Before Frozen Embryo Transfer
Acronym: SONTEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Massin Nathalie (Other)
Responsible Party: Sponsor-Investigator, Dr Massin Nathalie, Dr, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SONTEC
Record Dates: First submitted 2015-09-03; First posted 2016-07-15 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Fertility
Keywords: Ovulation Induction; quality of life; Reproductive Physiological Processes; fertility
MeSH Terms: interventions — Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural cycle (Other): Ovulation is not induced by drugs
  Interventions: Other: natural cycle
- Moderate ovarian stimulation (Experimental): Ovulation is induced by recombinant follitropin alpha and recombinant choriogonadotropin
  Interventions: Drug: moderate ovarian stimulation

INTERVENTIONS:
Other: natural cycle — Ovulation is not induced by drugs
  Other Names: natural
  Arms: Natural cycle
Drug: moderate ovarian stimulation — Ovulation is induced by recombinant follitropin alpha and recombinant choriogonadotropin
  Other Names: ovarian stimulation
  Arms: Moderate ovarian stimulation

SUMMARY:
Embryo freezing is a technique used regularly to optimize the pregnancy rate in case of infertility. This method is performed in presence of supernumerary embryo(s) after fresh transfer, or after freeze all embryos in case of medical reasons. It is necessary to control that the transfer is performed when the endometrium is receptive, which is essential for embryo implantation and pregnancy. This period is defined as the "implantation window". Endometrial preparation can be achieved by hormone replacement therapy (HRT) or moderate ovarian stimulation (SO). The implantation window can also be assessed by monitoring of a natural cycle (NC). The objectives of this open randomized study is to compare the number of visits (ultrasound and blood tests) induced by the SO or NC as well as the women quality of life in both groups.

DETAILED DESCRIPTION:
For infertile couples supported by in vitro fertilization, embryo freezing is a technique used regularly to optimize the pregnancy rate per retrieval of oocytes. This method is performed in case of supernumerary embryo(s) after fresh embryo transfer, or freeze all of the embryonic cohort in case of medical reasons preventing the transfer. The embryo or embryos can then be thawed and transferred (FET) to achieve a live birth. However, it is necessary to first ensure that the transfer is carried out at a time when the endometrium is receptive, which is essential for embryo implantation and pregnancy. This period is defined as the "implantation window". Endometrial preparation can be performed by hormone replacement therapy (HRT) or moderate ovarian stimulation (SO). The implantation window can also be assessed by the monitoring of a natural cycle (NC). The choice of the key moment for the transfer is determined by ovulation and / or the rise of progesterone. To date, no study has demonstrated the superiority of one protocol over another in terms of birth rates. In the investigative center, treatment is usually carried out by daily subcutaneous injections of gonadotrophins followed by ovulation induction. In this context, the implementation of the FET in natural cycle may appear less burdensome for the patient and more physiological. The consideration is additional constraints, NC imposing more frequent monitoring (ultrasound and / or hormone assays) to detect the ovulation peak and less freedom in choosing the date of transfer. The average number of visits with SO is 2.6 per cycle. The aim of this study is to compare the stresses and safety of these two therapeutic proposals to determine the least restrictive for patients.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to the general social security regime and benefiting from 100% infertility;
* Regular Cycles 26 to 35 days;
* Support in IVF or ICSI ;
* Existence of at least 2 frozen embryos to J2 or J3;
* Treated for their first or second cycle of TEC.

Exclusion Criteria:

* Donor sperm;
* Irregular cycles and / or polycystic ovary syndrome;
* Embryos frozen at J1 or J5 / J6 or double planned transfer or transfer of 3 embryos intended;
* Patients who have had more than 3 transfers or more than 6 embryos replaced without pregnancy or puncture rank> 3;
* uterine malformation existing;
* Presence of a hydrosalpinx.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of visits | From inclusion visit to embryo transfer : up to 90 days
  number of visits (for clinical examination, ultrasound and hormonal dosage) required to monitor ovulation in both groups

SECONDARY OUTCOMES:
Fertiqol | From inclusion visit to embryo transfer : up to 90 days
  the score of quality of life related to the couple's infertility, the Fertiqol questionnaire, a questionnaire validated by the European Society of Human Reproduction and Embryology (ESHRE) and taking into account the tolerance to treatment;
defrost cancellation rate | From inclusion visit to embryo transfer : up to 90 days
  the defrost cancellation rate cycle started, whatever the cause: Early ovulation problem of organization, ... excluding "non-transfer" related to embryo lysis thawing
transfer on weekends and holidays | From inclusion visit to embryo transfer : up to 90 days
  the transfer rate on weekends and holidays
HCG levels> 100 U / L | From inclusion visit to pregnancy test : up to 100 days
  the incipient pregnancy rate per transfer defined by a HCG levels> 100 U / L
pregnancy | From pregnancy test to ultrasound at 6 week of gestation : up to 100 days
  the rate of pregnancy by ultrasound transfer defined by the presence of a cardiac activity
Birth | From transfer to delivery : up to 9 months
  The live birth rate per transfer defined by the birth of at least one living child
Gestationnal age at delivery | From transfer to delivery : up to 9 months
  the term of delivery
Implantation | From transfer to delivery : up to 9 months
  the implantation rate defined by the total number of live births to the total number of embryos replaced
Miscarriage | From pregnancy test to ultrasound at 6 week of gestation : up to 100 days
  the rate of early miscarriage (before 12 SA)
Cost | From pregnancy test to ultrasound at 6 week of gestation : up to 100 days
  the average estimated cost of drug treatment and monitoring (ultrasound and hormone assays).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massin, MD, Principal Investigator — CHIC
Locations (1):
- CHI Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjuresten K, Landgren BM, Hovatta O, Stavreus-Evers A. Luteal phase progesterone increases live birth rate after frozen embryo transfer. Fertil Steril. 2011 Feb;95(2):534-7. doi: 10.1016/j.fertnstert.2010.05.019. Epub 2010 Jun 26. PMID 20579989
- [Background] Boivin J, Takefman J, Braverman A. The fertility quality of life (FertiQoL) tool: development and general psychometric properties. Hum Reprod. 2011 Aug;26(8):2084-91. doi: 10.1093/humrep/der171. Epub 2011 Jun 10. PMID 21665875
- [Background] de La Rochebrochard E, Quelen C, Peikrishvili R, Guibert J, Bouyer J. Long-term outcome of parenthood project during in vitro fertilization and after discontinuation of unsuccessful in vitro fertilization. Fertil Steril. 2009 Jul;92(1):149-56. doi: 10.1016/j.fertnstert.2008.05.067. Epub 2008 Aug 15. PMID 18706550
- [Background] Eftekhar M, Rahmani E, Pourmasumi S. Evaluation of clinical factors influencing pregnancy rate in frozen embryo transfer. Iran J Reprod Med. 2014 Jul;12(7):513-8. PMID 25114675
- [Background] El Bahja D, Hertz P, Schweitzer T, Lestrade F, Ragage JP. [Frozen embryo transfer protocol: does spontaneous cycle give good results?]. Gynecol Obstet Fertil. 2013 Nov;41(11):648-52. doi: 10.1016/j.gyobfe.2011.08.007. Epub 2012 Feb 16. French. PMID 22342107
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Background] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Background] Haouzi D, Assou S, Mahmoud K, Tondeur S, Reme T, Hedon B, De Vos J, Hamamah S. Gene expression profile of human endometrial receptivity: comparison between natural and stimulated cycles for the same patients. Hum Reprod. 2009 Jun;24(6):1436-45. doi: 10.1093/humrep/dep039. Epub 2009 Feb 26. PMID 19246470
- [Background] Nargund G, Wei CC. Successful planned delay of ovulation for one week with indomethacin. J Assist Reprod Genet. 1996 Sep;13(8):683-4. doi: 10.1007/BF02069650. No abstract available. PMID 8897131
- [Background] Park SJ, Goldsmith LT, Skurnick JH, Wojtczuk A, Weiss G. Characteristics of the urinary luteinizing hormone surge in young ovulatory women. Fertil Steril. 2007 Sep;88(3):684-90. doi: 10.1016/j.fertnstert.2007.01.045. Epub 2007 Apr 16. PMID 17434509
- [Background] Tobler KJ, Zhao Y, Weissman A, Majumdar A, Leong M, Shoham Z. Worldwide survey of IVF practices: trigger, retrieval and embryo transfer techniques. Arch Gynecol Obstet. 2014 Sep;290(3):561-8. doi: 10.1007/s00404-014-3232-6. Epub 2014 Apr 18. PMID 24744054
- [Background] Tomas C, Alsbjerg B, Martikainen H, Humaidan P. Pregnancy loss after frozen-embryo transfer--a comparison of three protocols. Fertil Steril. 2012 Nov;98(5):1165-9. doi: 10.1016/j.fertnstert.2012.07.1058. Epub 2012 Jul 27. PMID 22840239
- [Background] Troude P, Guibert J, Bouyer J, de La Rochebrochard E; DAIFI Group. Medical factors associated with early IVF discontinuation. Reprod Biomed Online. 2014 Mar;28(3):321-9. doi: 10.1016/j.rbmo.2013.10.018. Epub 2013 Oct 31. PMID 24461478
- [Background] Weissman A, Levin D, Ravhon A, Eran H, Golan A, Levran D. What is the preferred method for timing natural cycle frozen-thawed embryo transfer? Reprod Biomed Online. 2009 Jul;19(1):66-71. doi: 10.1016/s1472-6483(10)60048-x. PMID 19573293
- [Background] Yu J, Ma Y, Wu Z, Li Y, Tang L, Li Y, Deng B. Endometrial preparation protocol of the frozen-thawed embryo transfer in patients with polycystic ovary syndrome. Arch Gynecol Obstet. 2015 Jan;291(1):201-11. doi: 10.1007/s00404-014-3396-0. Epub 2014 Jul 31. PMID 25091221